CLINICAL TRIAL: NCT07006727
Title: A Phase I, Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Dosimetry, and Preliminary Activity of [225Ac]Ac-ETN029 in Patients With Advanced DLL3-expressing Solid Tumors
Brief Title: Phase I Study of [225Ac]Ac-ETN029 in Patients With Advanced DLL3-expressing Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CESP359A12101; 2024-519111-34-00 (Other: EU CTIS number)
Record Dates: First submitted 2025-05-16; First posted 2025-06-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Carcinoma; Large Cell Neuroendocrine Carcinoma of the Lung; Neuroendocrine Prostate Cancer; Gastroenteropancreatic Neuroendocrine Carcinoma
Keywords: Small Cell Lung Carcinoma (SCLC); Large Cell Neuroendocrine Carcinoma of the Lung (LCNEC); Neuroendocrine Prostate Cancer (NEPC); Gastroenteropancreatic Neuroendocrine Carcinoma (GEP-NEC); DLL3; Neuroendocrine neoplasms; Radioligand therapy (RLT); [225Ac]Ac-ETN029; [111In]In-ETN029
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive 225Ac-ETN029, with some patients also receiving 111In-ETN029
  Interventions: Drug: 225Ac-ETN029; Drug: 111In-ETN029

INTERVENTIONS:
Drug: 225Ac-ETN029 — Radioligand therapy
Drug: 111In-ETN029 — Radioligand imaging agent

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, dosimetry and preliminary efficacy of [225Ac]Ac-ETN029 and the safety and imaging properties of [111In]In-ETN029 in patients aged ≥ 18 years with locally advanced or metastatic DLL3 positive cancers.

DETAILED DESCRIPTION:
This is a phase I, open-label, multi-center study to evaluate the safety, tolerability, dosimetry, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of 225Ac-ETN029 in patients with advanced DLL3-expressing solid tumors. The study consists of a dose escalation part, followed by a dose expansion part. Once the recommended radioactive dose(s) of 225Ac-ETN029 for further clinical evaluation are determined, the dose expansion part will further characterize the safety, tolerability, and preliminary anti-tumor activity of 225Ac-ETN029. The study will also enable an initial evaluation of the safety, dosimetry, PK, and imaging properties of 111In-ETN029.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients with one of the following indications:
* Locally advanced, unresectable, or metastatic SCLC with disease progression following, or intolerance to, at least 1 line of systemic therapy, including platinum-containing chemotherapy, unless patient was ineligible to receive such therapy. Prior DLL3-targeted therapy is allowed. For dose expansion, patients should have received no more than 2 prior lines of systemic therapy.
* Dose escalation only: LCNEC of the lung with disease progression following, or intolerance to, at least 1 line of systemic therapy, including platinum-containing chemotherapy, unless patient was ineligible to receive such therapy.
* Dose expansion only: Locally advanced, unresectable, or metastatic de novo or castration-resistant, treatment-emergent NEPC with neuroendocrine differentiation confirmed by local histology and NEPC marker expression (e.g., chromogranin, synaptophysin) confirmed by local IHC. Prior PSMA-targeted, Lu-177-based RLT is allowed. Patients must have at least one measurable lesion (per RECIST 1.1) that shows 111In-ETN029 uptake higher than surrounding tissues on SPECT/CT as assessed by the Investigator.
* Dose expansion only: Locally advanced, unresectable, or metastatic GEP-NEC with disease progression following, or intolerance to, at least 1 line of systemic therapy, including platinum-containing chemotherapy, unless patient was ineligible to receive such therapy. Patients must have at least one measurable lesion (per RECIST 1.1) that shows 111In-ETN029 uptake higher than surrounding tissues on SPECT/CT as assessed by the Investigator.

Exclusion Criteria:

* Absolute neutrophil count (ANC) < 1.0 x 109/L, hemoglobin < 9 g/dL, or platelet count < 75 x 109/L
* QT interval corrected by Fridericia's formula (QTcF) ≥ 470 msec
* eGFR < 60 mL/min (<0.835 mL/s), calculated using the CKD-EPI 2021 formula or measured
* Unmanageable urinary tract obstruction or urinary incontinence
* Presence of leptomeningeal disease, of symptomatic CNS metastases or of CNS metastases that require local CNS-directed therapy
* History of or current interstitial lung disease or pneumonitis ≥ Grade 2
* Any prior DLL3-targeted therapy (except for SCLC) and any prior RLT (except for NEPC)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2031-06-17 (Estimated); Study Completion 2031-06-17 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities of 225Ac-ETN029 | From the start of study treatment until 6 weeks after
  A dose limiting toxicity (DLT) is defined as any adverse event or abnormal laboratory value of CTCAE 5.0 grade 3 or higher that occurs within the DLT evaluation period and that is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications with a few exceptions defined in the study protocol. Other significant toxicities may be considered to be DLTs, even if not Grade 3 or higher.
Incidence and severity of adverse events and serious adverse events of 225Ac-ETN029 | From start of study treatment until completion of the 36 month follow up, assessed up to approximately 42 months
  Incidence and severity of treatment-emergent adverse events and serious adverse events, including changes in laboratory values, vital signs, and electrocardiograms qualifying and reported as AEs
Dose modifications for 225Ac-ETN029 | From the start of study treatment until last dose of study treatment, assessed as approximately 24 weeks
  Number of dose modifications (e.g, dose interruptions and reductions) for 225Ac-ETN029
Dose intensity for 225Ac-ETN029 | From start of study treatment until last dose of study treatment, assessed as approximately 24 weeks
  Dose intensity of 225Ac-ETN029 defined as the ratio of actual cumulative dose received and actual duration of exposure

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 42 months
  ORR is defined as the proportion of patients with a BOR of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines.
Disease control rate (DCR) | Up to approximately 42 months
  DCR is defined as the proportion of patients with a BOR of CR, PR, or stable disease according to RECIST v1.1 guidelines.
Duration of response (DOR) | Up to approximately 42 months
  DOR is defined as the time between the first documented response (CR or PR) and the date of progression according to RECIST v1.1 guidelines, or death due to any cause.
Progression free survival (PFS) | Up to approximately 42 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression according to RECIST v1.1 guidelines or death due to any cause.
Area under the curve (AUC) of 225Ac-ETN029 and 111In-ETN029 | During the first ~14 days following 225Ac-ETN029 administration and ~5 days following 111In-ETN029 administration
  Area under the concentration time curve. AUC is a PK parameter that will be determined using non-compartmental analysis (NCA).
Observed maximum blood concentration (Cmax) of 225Ac-ETN029 and 111In-ETN029 | During the first ~14 days following 225Ac-ETN029 administration and ~5 days following 111In-ETN029 administration
  The maximum (peak) observed blood drug concentration after single dose administration. Cmax is a PK parameter that will be determined using non-compartmental analysis (NCA).
Volume of distribution (Vz) of 225Ac-ETN029 and 111In-ETN029 during the terminal phase | During the first ~14 days following 225Ac-ETN029 administration and ~5 days following 111In-ETN029 administration
  The apparent volume of distribution during terminal phase. Vz is a PK parameter that will be determined using non-compartmental analysis (NCA).
Terminal elimination half-life (T1/2) of 225Ac-ETN029 and 111In-ETN029 | During the first ~14 days following 225Ac-ETN029 administration and ~5 days following 111In-ETN029 administration
  The elimination half-life associated with the terminal slope of a semi logarithmic concentration-time curve. T1/2 (associated with a terminal slope) is a PK parameter that will be determined using non-compartmental analysis (NCA).
Total body clearance of 225Ac-ETN029 and 111In-ETN029 | During the first ~14 days following 225Ac-ETN029 administration and ~5 days following 111In-ETN029 administration
  The total body clearance of drug from the plasma. Clearance is a PK parameter that will be determined using non-compartmental analysis (NCA).
Observed maximum radioactivity concentration (Rmax) of 225Ac-ETN029 | During the first ~14 days following 225Ac-ETN029 administration and ~5 days following 111In-ETN029 administration
  The maximum (peak) observed blood radioactivity concentration after single dose administration. Rmax is a PK parameter that will be determined using non-compartmental analysis (NCA).
Absorbed dose of 225Ac-ETN029 and 111In-ETN029 | During the first ~14 days following 225Ac-ETN029 administration and ~5 days following 111In-ETN029 administration
  The absorbed dose will be determined based on time activity curves (TACs) obtained from the radiotracer uptake (as percentage of injected dose) via quantification of images.
Incidence and severity of adverse events and serious adverse events of 111In-ETN029 | From the start of 111In-ETN029 to the day before the first 225Ac-ETN029 administration or until the completion of 30 day follow up (assessed as approximately 30 days)
  Incidence and severity of treatment-emergent adverse events and serious adverse events
Visual and quantitative assessment of 111In-ETN029 uptake in normal tissues over time | During the first ~5 days following 111In-ETN029 administration
  Quantitative assessment expressed as standardized uptake values (SUVs) of 111In-ETN029 uptake in normal tissues

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - University Of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.